CLINICAL TRIAL: NCT02394145
Title: The Relationship Between Genotype and Platelet Reactivity in Patients Treated With Ticagrelor Versus Clopidogrel: PIANO Genotype Study
Brief Title: Genotype and Platelet Reactivity in Patients on Hemodialysis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Weon Kim, Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PIANO-genetics
Record Dates: First submitted 2015-03-14; First posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Kidney Disease
Keywords: platelet; ticagrelor; clopidogrel; end stage renal disease; hemodialysis; genetics
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Ticagrelor 180mg in ESRD patients (Experimental): After randomization, ESRD patients on HD will be treated by an initial loading dose of ticagrelor (180 mg) and maintenance doses (ticagrelor 90 mg twice daily) for 14 days. Platelet reactivity and genetic polymorphism will be assessed.
  Interventions: Drug: Ticagrelor
- Clopidogrel 75mg in ESRD patients (Active Comparator): After randomization, ESRD patients on HD will be treated by an initial loading dose of clopidogrel 300 mg) and maintenance doses (clopidogrel 75 mg once a day) for 14 days. Platelet reactivity and genetic polymorphism will be assessed.
  Interventions: Drug: Clopidogrel
- Clopidogrel 150mg in ESRD patients (Active Comparator): After randomization, ESRD patients on HD will be treated by an initial loading dose of clopidogrel 300 mg) and maintenance doses (clopidogrel 150 mg once a day) for 14 days. Platelet reactivity and genetic polymorphism will be assessed.
  Interventions: Drug: Clopidogrel
- Ticagrelor 180mg in normal kidney (Active Comparator): After randomization, patients with normal kidney function will be treated by an initial loading dose of ticagrelor (180 mg) and maintenance doses (ticagrelor 90 mg twice daily) for 14 days. Platelet reactivity and genetic polymorphism will be assessed
  Interventions: Drug: Ticagrelor
- Clopidogrel 75mg in normal kidney (Active Comparator): After randomization, patients with normal kidney function will be treated by an initial loading dose of clopidogrel 300 mg) and maintenance doses (clopidogrel 75 mg once a day) for 14 days. Platelet reactivity and genetic polymorphism will be assessed.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Patients with normal kidney function and ESRD on hemodialysis will be treated by ticagrelor 90mg twice a day for 14 days. After then, platelet reactivity will be assessed by light aggregometry and VerifyNow assay.
  Other Names: Brilinta
  Arms: Ticagrelor 180mg in ESRD patients; Ticagrelor 180mg in normal kidney
Drug: Clopidogrel — Patients with normal kidney function and ESRD on hemodialysis will be treated by clopidogrel 75mg or 150mg once a day for 14 days. After then, platelet reactivity will be assessed by light aggregometry and VerifyNow assay.
  Other Names: Plavix
  Arms: Clopidogrel 150mg in ESRD patients; Clopidogrel 75mg in ESRD patients; Clopidogrel 75mg in normal kidney

SUMMARY:
Patients with end stage renal disease (ESRD) on hemodialysis (HD) exhibited higher platelet reactivity to clopidogrel than did those with normal renal function. We recently reported platelet inhibition by ticagrelor was faster and markedly greater than by clopidogrel with onset dosing regimen in patients with ESRD on HD. However, few studies have been conducted genetic influence in high platelet reactivity in patients with ESRD on HD.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a strong risk factor for cardiovascular morbidity and mortality, and confers an increasing risk of stent thrombosis even when dual antiplatelet therapy (clopidogrel and aspirin) is administered. Patients with severe CKD or end stage renal disease (ESRD) on hemodialysis (HD) exhibited higher platelet reactivity to clopidogrel than did those with normal renal function. We recently reported platelet inhibition by ticagrelor was markedly greater than by clopidogrel in patients with ESRD on HD. But exact mechanism of high platelet reactivity in ESRD patients was not fully evaluated. A possible postulation would be genetic influence. To investigate this issue, we will evaluate genetic polymorphism in patients with normal kidney function and ESRD on HD according to different doses of clopidogrel and ticagrelor. Genetic test will be assessed polymorphism of ABCB1, PON1, CYP2C19, CYP2C9 and P2Y12.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients undergoing regular (≥ 6 months) maintenance HD
* Matching patients with normal kidney function
* documented coronary artery disease or high risk (Framingham heart risk score ≥ 20%) of coronary artery disease

Exclusion Criteria:

* known allergies to aspirin, clopidogrel, or ticagrelor
* concomitant use of other antithrombotic drugs (oral anticoagulants, dipyridamole)
* thrombocytopenia (platelet count <100,000/mm3)
* hematocrit <25%
* uncontrolled hyperglycemia (hemoglobin A1c >10%)
* liver disease (bilirubin level >2 mg/dl)
* symptomatic severe pulmonary disease
* active bleeding or bleeding diathesis
* gastrointestinal bleeding within the last 6 months
* hemodynamic instability
* acute coronary or cerebrovascular event within the last 3 months
* pregnancy
* any malignancy
* concomitant use of a cytochrome P450 inhibitor or nonsteroidal anti-inflammatory drug
* recent treatment (<30 days) with a glycoprotein IIb/IIIa antagonist

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
The difference of antiplatelet effects according to genotype | 14 days after study drug treatment
  The difference of P2Y12 reaction units (PRUs) according to genotype

SECONDARY OUTCOMES:
The difference of antiplatelet effects according to kidney function | 14 days after study drug treatment
  The difference of P2Y12 reaction units (PRUs) according to kidney function

CONTACTS AND LOCATIONS:
Overall Officials: Weon Kim, MD, PhD, Principal Investigator — Kyung Hee University Hospital
Locations (1):
- Kyung Hee University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730